CLINICAL TRIAL: NCT06001970
Title: Activity Pacing, Fatigue Management, and Self-regulation Strategies as a Promising Approach for Managing Fatigue Symptoms and for Promoting Physical Activity in Adults Who Experience Fatigue
Brief Title: Activity Pacing for Fatigue Management
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Northumbria University (Other)
Collaborators: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 313465
Record Dates: First submitted 2023-05-05; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Fatigue; Chronic Condition; Self-regulation; Physical Activity; Activity Pacing
Keywords: physical activity behavior; self-regulation; fatigue; chronic condition
MeSH Terms: conditions — Fatigue; Chronic Disease; Self-Control; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Adults who experience fatigue and have been through an activity pacing program: Adults with chronic conditions who experience fatigue recruited from Cresta Fatigue Clinic, Newcastle, UK
- Adults who experience fatigue and have not been through an activity pacing program: Adults with chronic conditions who experience fatigue recruited from the waiting list of Cresta Fatigue Clinic, Newcastle, UK
- Health professionals working on activity pacing: Health professionals who are working on Cresta Fatigue Clinic, Newcastle, UK

SUMMARY:
This project will focus on perceived fatigue as a barrier to physical activity participation and will explore if and how activity pacing, fatigue management, and self-regulation strategies can help to overcome this barrier in adults with chronic conditions who experience fatigue symptoms. The main aims are:

1. To demonstrate the differences and similarities on activity pacing, perceived fatigue, self-regulation, physical activity, and health-related quality of life in adults who experience fatigue by comparing individuals who have been through an activity pacing program or not.
2. To explore thoughts, experiences, needs, and perspectives on activity pacing of adults with fatigue and health professionals as well as any ideas for future development of an optimal intervention.

Participants will be invited to complete questionnaires on several variables (activity pacing, physical activity, fatigue, health-related quality of life, and self-regulation of physical activity). In addition, they will be invited to wear an Actigraph for 7 full days and they will also be invited to a focus group interview.

DETAILED DESCRIPTION:
Activity pacing is a fatigue management strategy that regulates energy and activity levels while maintaining or increasing engagement in physical activity. This approach is particularly beneficial for individuals with chronic conditions who experience significant fatigue as they often struggle with sustained physical activity participation due to recurring patterns of overexertion and subsequent fatigue or pain. Therefore, activity pacing strategies are important because individuals learn to manage fatigue symptoms, optimize physical activity behaviour, and accomplish a more stable activity pacing pattern, which will improve their health-related quality of life and well-being.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a chronic condition
* Experience fatigue
* Ambulatory

Exclusion Criteria:

* Children
* Wheelchair users

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with chronic conditions who experience fatigue
Sampling Method: Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Perceived fatigue | 1 point in time measuring for the past 7 days
  Fatigue Severity Scale is a 9-item questionnaire assessing the impact of perceived fatigue in adults with chronic disorders. FSS is valid and reliable to determine the impact of perceived fatigue among several clinical populations.
Physical activity | 1 point in time measuring for the past 7 days
  Self-reported PA: IPAQ is a 7-item measure that assesses the intensity of physical activity and sitting time in their daily lives . It has been validated in adults with stroke .
Engagement in Pacing and Perceived Risk of Overactivity | 1 point in time measuring for the past 7 days
  The Activity Pacing Questionnaire (APQ) is a 7-item measure assessing activity pacing and risk of overactivity. Reliability and construct validity have been investigated and the paper is in preparation.
Perceived Fatigue | 1 point in time measuring for the past 7 days
  2)FACIT-F (version 4) is a 40-item questionnaire evaluating self-reported fatigue and its influence on everyday activities and function among adults with cancer and older people experiencing fatigue . FACIT-F is valid and reliable in several patient populations.
Objective Physical Activity | 7 days
  Participants will be invited to wear an Actigraph for 7 full days.

SECONDARY OUTCOMES:
Self-regulation | 1 point in time measuring for the past 7 days
  Physical Activity Self-Regulation scale (PASR-12) is a 12-item measure assessing self-regulation for physical activity. PASR-12 has demonstrated validity and reliability in older adults.
Health-related Quality of Life | 1 point in time measuring for the past 7 days
  RAND-12 health status inventory is a 12-item questionnaire that evaluates the health-related quality of life. Literature supports acceptable construct validity and test-retest reliability of the RAND-12 among clinical populations.

CONTACTS AND LOCATIONS:
Locations (1):
- Northumbria University, Newcastle, United Kingdom